CLINICAL TRIAL: NCT00716443
Title: Open-Label, Randomized, Split-Face Study to Evaluate the Efficacy, Safety and Subject Satisfaction of Pain Management During and After Restylane® Dermal Filler Injections for the Correction of Nasolabial Folds
Brief Title: Evaluate Efficacy, Safety & Subject Satisfaction of Pain Management With Pliaglis® Cream for Dermal Filler Injections
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: US10098
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Results first posted 2010-02-01 (Estimated); Last update posted 2022-08-23 (Actual); Status verified 2012-09

CONDITIONS: Nasolabial Folds
Keywords: Nasolabial folds; wrinkles; topical anesthetic
MeSH Terms: interventions — Tetracaine; Lidocaine; Benzocaine; Ointments

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pliaglis® Cream (Active Comparator): tetracaine 4% / lidocaine 7% cream; this was a randomized, split face study where Pliaglis® Cream was used on one side of the face and a compounded topical anesthetic ointment was used on the other side of the face. Restylane® was injected into both sides of the face.
  Interventions: Drug: tetracaine 7% / lidocaine 7% cream (Pliaglis® Cream); Drug: benzocaine 20% / lidocaine 6% / tetracaine 4% ointment
- benzocaine 20% / lidocaine 6% / tetracaine 4% ointment (Active Comparator): apply benzocaine / lidocaine / tetracaine ointment once on the other side of the face prior to Restylane® injections; this was a randomized, split face study where Pliaglis® Cream was used on one side of the face and a compounded topical anesthetic ointment was used on the other side of the face. Restylane® was injected into both sides of the face.
  Interventions: Drug: benzocaine 20% / lidocaine 6% / tetracaine 4% ointment

INTERVENTIONS:
Drug: tetracaine 7% / lidocaine 7% cream (Pliaglis® Cream) — Apply tetracaine/lidocaine cream once on one side of the face prior to Restylane® injections
  Other Names: Pliaglis® Cream
  Arms: Pliaglis® Cream
Drug: benzocaine 20% / lidocaine 6% / tetracaine 4% ointment — apply benzocaine / lidocaine / tetracaine ointment once on the other side of the face prior to Restylane® injections
  Other Names: BLT ointment

SUMMARY:
Pliaglis® Cream versus compounded topical anesthetic for pain management during Restylane® injections for the correction of nasolabial folds.

DETAILED DESCRIPTION:
Open-label, randomized study designed to assess the effectiveness of a topical anesthetic (Pliaglis® Cream) versus a compounded topical anesthetic at needle stick, immediately after, one and three hours after Restylane® injections in the nasolabial folds.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female Subjects 30 - 65 years of age
* Subject undergoing cosmetic dermal filler injections for correction of nasolabial folds. Treatment sites should be comparable, requiring the same number of injections on each nasolabial fold
* Subjects diagnosed with moderate nasolabial folds (Wrinkle Severity Rating Scale of grade 3)

Exclusion Criteria:

* Subjects under treatment for a dermatologic condition on the face, which may interfere with the safe evaluation of the study treatment (e.g. eczema, psoriasis, severe sun-damage, dermatitis), have damaged, denuded or broken skin at the designated treatment site and/or have scarring or infection of the area to be treated
* Subjects who have taken prescription or non-prescription analgesic medication during the 24 hour period prior to the procedure
* Subjects with a history of bleeding or clotting disorders
* Subjects who have used ASA (aspirin), NSAIDs (Non-Steroidal Anti- inflammatory Drugs), anticoagulants, St. John's Wort or high doses of Vitamin E (above the recommended daily allowance) within 2 weeks prior to the procedure

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald W Gottschalk, MD, Study Director — Galderma R&D
Locations (4):
- United States (4):
  - Skin and Cancer Associates, Center for Cosmetic Enhancement, Aventura, Florida
  - Palm Beach Esthetic Dermatology and Laser Center, West Palm Beach, Florida
  - Sadick Dermatology, New York, New York
  - Premier Clinical Research, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period: First subject was enrolled on July 30, 2008 and the last subject was enrolled on September 8, 2008.
Pre-assignment Details: The wash-out period prior to baseline was 24 hrs for analgesic medication; 14 days for aspirin (ASA), non-steroidal anti-inflammatory drugs (NSAIDs), anticoagulants, St. John's Wort or doses of Vitamin E above the recommended daily allowance; 14 days for sunburn/tanning bed exposure; 12 months for filler injections into the nasolabial folds.
Groups:
- Pliaglis® Cream and Compounded Topical Anesthetic Ointment: Apply Pliaglis® Cream on one side of the face and compounded topical anesthetic ointment on the other side of the face; this was a randomized, split face study where Pliaglis® Cream was used on one side of the face and compounded topical anesthetic ointment was used on the other side of the face prior to injection of Restylane® into the nasolabial folds.
Period: Overall Study
Arm/Group | Pliaglis® Cream and Compounded Topical Anesthetic Ointment
Started | 51
Completed | 51
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pliaglis® Cream and Compounded Topical Anesthetic Ointment
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (8.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Subject's Pain Evaluation by Visual Analog Scale (VAS)Upon First Needlestick, Immediately After Injection, One Hour After Injection and Three Hours After Injection of Restylane® Into the Nasolabial Folds
Description: Subject's pain as evaluated using a VAS scale from 0 - 10 cm (centimeters) with 0 cm being no pain and 10 cm being the worst pain imaginable upon first needlestick, immediately after injection, one hour after injection and three hours after injection of Restylane® into the nasolabial folds
Time Frame: upon first needlestick, immediately after injection, one hour after injection and three hours after injection of Restylane® into the nasolabial folds
Population: ITT (Intent to Treat), LOCF (Last Observation Carried Forward)
Measure: Mean (Standard Deviation); unit: centimeters
Groups:
- Pliaglis® Cream: Pliaglis® Cream
- Compounded Topical Anesthetic Ointment: compounded topical anesthetic ointment
Arm/Group | Pliaglis® Cream | Compounded Topical Anesthetic Ointment
Number analyzed (Participants) | 51 | 51
centimeters
  upon first needle stick | 2.3 (2.07) | 2.8 (2.17)
  immediately after injection | 2.7 (2.14) | 2.8 (2.22)
  one hour after injection | 0.8 (1.12) | 0.6 (0.93)
  three hours after injection | 0.5 (1.14) | 0.5 (0.91)

2. Secondary Outcome: Number of Participants Who Answered the Question "What Level of Pain Did You Experience When You Were Injected?" Three Hours After Injection of Restylane® Into the Nasolabial Folds
Description: Number of participants who answered according to a scale of None, Minimal, Mild, Moderate, Severe, or No response to the question "What level of pain did you experience when you were injected?" three hours after injection of Restylane® into the nasolabial folds
Time Frame: three hours after injection of Restylane® into the nasolabial folds
Population: ITT (Intent to Treat), LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Arm/Group | Pliaglis® Cream | Compounded Topical Anesthetic Ointment
Number analyzed (Participants) | 51 | 51
participants
  None | 4 | 2
  Minimal | 23 | 24
  Mild | 15 | 15
  Moderate | 8 | 9
  Severe | 1 | 1
  No response | 0 | 0

3. Secondary Outcome: Number of Participants Who Answered the Question "If You Experienced Pain, Was it What You Expected From the Injection Procedure?" Three Hours After Injection of Restylane® Into the Nasolabial Folds
Description: Number of participants who answered No, Yes, Had no expectations or No response to the question "If you experienced pain, was it what you expected from the injection procedure?" three hours after injection of Restylane® into the nasolabial folds
Time Frame: three hours after injection of Restylane® into the nasolabial folds
Population: ITT (Intent to Treat), LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Arm/Group | Pliaglis® Cream | Compounded Topical Anesthetic Ointment
Number analyzed (Participants) | 51 | 51
participants
  No | 10 | 8
  Yes | 27 | 29
  Had no expectations | 12 | 13
  No response | 2 | 1

4. Secondary Outcome: Number of Participants Who Answered the Question "If it Was Different Than What You Expected, Was it?" Three Hours After Injection of Restylane® Into the Nasolabial Folds
Description: Number of participants who answered the question "If it was different than what you expected, was it?" (More pain, Less pain or No response) three hours after injection of Restylane® into the nasolabial folds
Time Frame: three hours after injection of Restylane® into the nasolabial folds
Population: ITT (Intent to Treat), LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Arm/Group | Pliaglis® Cream | Compounded Topical Anesthetic Ointment
Number analyzed (Participants) | 51 | 51
participants
  More pain | 10 | 9
  Less pain | 14 | 14
  No response | 27 | 28

5. Secondary Outcome: Number of Participants Who Answered the Question "Still Speaking to the Topical Anesthetic You Had on the Right/Left Side of Your Face, Would You Recommend it to Your Friend or Family Member?" 3 Hours After Injection of Restylane® Into Nasolabial Folds
Description: Number of participants who answered No, Yes or No response to the question "Still speaking to the topical anesthetic you had on the right/left side of your face, would you recommend it to your friend or family member?" three hours after injection of Restylane® into the nasolabial folds
Time Frame: three hours after injection of Restylane® into the nasolabial folds
Population: ITT (Intent to Treat), LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Arm/Group | Pliaglis® Cream | Compounded Topical Anesthetic Ointment
Number analyzed (Participants) | 51 | 51
participants
  No | 13 | 12
  Yes | 38 | 39
  No response | 0 | 0

6. Secondary Outcome: Number of Participants in Each Category of the Investigator Evaluation of the Subject's Post Procedure Pain Assessment Scale Upon First Needle Stick of Injection of Restylane® Into the Nasolabial Folds
Description: Number of participants in each category of the Investigator Evaluation of the Subject's Post Procedure Pain Assessment scale (0 = No pain; 1 = Slight pain; 2 = Moderate pain; 3 = Severe pain) upon first needle stick of an injection of Restylane® into the nasolabial folds
Time Frame: Upon first needle stick of injection of Restylane® into the nasolabial folds
Population: ITT (Intent to Treat), LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Arm/Group | Pliaglis® Cream | Compounded Topical Anesthetic Ointment
Number analyzed (Participants) | 51 | 51
participants
  No pain | 17 | 13
  Slight pain | 28 | 25
  Moderate pain | 6 | 12
  Severe pain | 0 | 1

7. Secondary Outcome: Number of Participants in Each Category of the Investigator Evaluation of the Subject's Post Procedure Pain Assessment Scale Immediately After Injection of Restylane® Into the Nasolabial Folds
Description: Number of participants in each category of the Investigator Evaluation of the Subject's Post Procedure Pain Assessment scale (0 = No pain; 1 = Slight pain; 2 = Moderate pain; 3 = Severe pain) immediately after injection of Restylane® into the nasolabial folds immediately after injection of Restylane® into the nasolabial folds
Time Frame: immediately after injection of Restylane® into the nasolabial folds
Population: ITT (Intent to Treat), LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Arm/Group | Pliaglis® Cream | Compounded Topical Anesthetic Ointment
Number analyzed (Participants) | 51 | 51
participants
  No pain | 35 | 29
  Slight pain | 10 | 15
  Moderate pain | 6 | 7
  Severe pain | 0 | 0

8. Secondary Outcome: Number of Participants in Each Category of the Investigator's Evaluation of Subject's Pain Scale One Hour After Injection of Restylane® Into the Nasolabial Folds
Description: Number of participants in each category of the Investigator's Evaluation of Subject's Pain scale (0 = No pain; 1 = Slight pain; 2 = Moderate pain; 3 = Severe pain) one hour after injection of Restylane® into the nasolabial folds
Time Frame: one hour after injection of Restylane® into the nasolabial folds
Population: ITT (Intent to Treat), LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Arm/Group | Pliaglis® Cream | Compounded Topical Anesthetic Ointment
Number analyzed (Participants) | 51 | 51
participants
  No pain | 49 | 49
  Slight pain | 2 | 2
  Moderate pain | 0 | 0
  Severe pain | 0 | 0

9. Secondary Outcome: Number of Participants in Each Category of the Investigator's Evaluation of Subject's Pain Scale Three Hours After Injection of Restylane® Into the Nasolabial Folds
Description: Number of participants in each category of the Investigator's Evaluation of Subject's Pain scale (0 = No pain; 1 = Slight pain; 2 = Moderate pain; 3 = Severe pain) three hours after injection of Restylane® into the nasolabial folds
Time Frame: three hours after injection of Restylane® into the nasolabial folds
Population: ITT (Intent to Treat), LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Arm/Group | Pliaglis® Cream | Compounded Topical Anesthetic Ointment
Number analyzed (Participants) | 51 | 51
participants
  No pain | 50 | 49
  Mild pain | 1 | 2
  Moderate pain | 0 | 0
  Severe pain | 0 | 0

10. Secondary Outcome: Number of Participants in Each Category of the Blinded Evaluator's Evaluation of Subject's Pain Scale Upon First Needle Stick of Injection of Restylane® Into the Nasolabial Folds
Description: Number of participants in each category of the Blinded Evaluator's Evaluation of Subject's Pain scale (0 = No pain; 1 = Slight pain; 2 = Moderate pain; 3 = Severe pain) upon first needle stick of an injection of Restylane® into the nasolabial folds
Time Frame: upon first needle stick of injection of Restylane® into the nasolabial folds
Population: ITT (Intent to Treat), LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Arm/Group | Pliaglis® Cream | Compounded Topical Anesthetic Ointment
Number analyzed (Participants) | 51 | 51
participants
  No pain | 14 | 9
  Mild pain | 31 | 29
  Moderate pain | 6 | 13
  Severe pain | 0 | 0

11. Secondary Outcome: Number of Participants in Each Category of the Blinded Evaluator's Evaluation of Subject's Pain Scale Immediately After Injection of Restylane® Into the Nasolabial Folds
Description: Number of participants in each category of the Blinded Evaluator's Evaluation of Subject's Pain scale (0 = No pain; 1 = Slight pain; 2 = Moderate pain; 3 = Severe pain) immediately after injection of Restylane® into the nasolabial folds
Time Frame: immediately after injection of Restylane® into the nasolabial folds
Population: ITT (Intent to Treat), LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Arm/Group | Pliaglis® Cream | Compounded Topical Anesthetic Ointment
Number analyzed (Participants) | 51 | 51
participants
  No pain | 35 | 28
  Slight pain | 11 | 18
  Moderate pain | 5 | 4
  Severe pain | 0 | 1

12. Secondary Outcome: Number of Participants in Each Category of the Blinded Evaluator's Evaluation of Subject's Pain Scale One Hour After Injection of Restylane® Into the Nasolabial Folds
Description: Number of participants in each category of the Blinded Evaluator's Evaluation of Subject's Pain scale (0 = No pain; 1 = Slight pain; 2 = Moderate pain; 3 = Severe pain) one hour after an injection of Restylane® into the nasolabial folds
Time Frame: one hour after injection of Restylane® into the nasolabial folds
Population: ITT (Intent to Treat), LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Arm/Group | Pliaglis® Cream | Compounded Topical Anesthetic Ointment
Number analyzed (Participants) | 51 | 51
participants
  No pain | 49 | 49
  Slight pain | 2 | 2
  Moderate pain | 0 | 0
  Severe pain | 0 | 0

13. Secondary Outcome: Number of Participants in Each Category of the Blinded Evaluator's Evaluation of Subject's Pain Scale Three Hours After Injection of Restylane® Into the Nasolabial Folds
Description: Number of participants in each category of the Blinded Evaluator's Evaluation of Subject's Pain scale (0 = No pain; 1 = Slight pain; 2 = Moderate pain; 3 = Severe pain) three hours after injection of Restylane® into the nasolabial folds
Time Frame: three hours after injection of Restylane® into the nasolabial folds
Population: ITT (Intent to Treat), LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Arm/Group | Pliaglis® Cream | Compounded Topical Anesthetic Ointment
Number analyzed (Participants) | 51 | 51
participants
  No pain | 50 | 50
  Mild pain | 1 | 1
  Moderate pain | 0 | 0
  Severe pain | 0 | 0

14. Secondary Outcome: Number of Participants With Yes/no Answers to Question to Investigator "Did the Topical Anesthetics Provide Adequate Anesthesia for the Injections of Restylane® Into the Nasolabial Folds Procedure?" Day of Injection of Restylane® Into Nasolabial Folds
Description: Number of participants with yes or no answers to question asked to investigator on the day of injection of Restylane® into the nasolabial folds "Did the topical anesthetics provided adequate anesthesia for the injections of Restylane® into the nasolabial folds procedure?"
Time Frame: Day of injection of Restylane® into the nasolabial folds
Population: ITT (Intent to Treat), LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Arm/Group | Pliaglis® Cream | Compounded Topical Anesthetic Ointment
Number analyzed (Participants) | 51 | 51
participants
  Yes | 44 | 44
  No | 7 | 7

15. Secondary Outcome: Number of Participants With Tolerability Assessments Resulting in Adverse Events From Baseline to Two Days After Injection of Restylane® Into the Nasolabial Folds
Description: Number of participants w/ tolerability assessments (erythema, edema, blanching) resulting in adverse events from Baseline to two days after injection of Restylane® into the nasolabial folds
Time Frame: Baseline to two days after injection of Restylane® into the nasolabial folds
Population: Safety
Measure: Number; unit: participants
Arm/Group | Pliaglis® Cream | Compounded Topical Anesthetic Ointment
Number analyzed (Participants) | 51 | 51
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to two days after Restylane® injections
Description: Subjects were asked if there had been any change in their health at each study visit; information obtained was recorded as adverse event9s), if applicable.
Arm/Group | Pliaglis® Cream and Compounded Topical Anesthetic Ointment
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 3/51
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pliaglis® Cream and Compounded Topical Anesthetic Ointment (N=51)
Implant site bruising (General disorders) | 3 (3) — Bruising is at Restylane® injection site

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigator has the right to publish or present the data resulting from this study, with agreed upon reviews by all interested parties, and in accordance with any confidentiality agreements that may exist.